CLINICAL TRIAL: NCT06595264
Title: Patients With Aneurysms of the Vein of Galen, H.U.B Experience; a Retrospective Study
Brief Title: Vein of Galen Aneurysm
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2024207
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Vein of Galen Malformation
Keywords: vein of Galen aneurysm; neuroradiological embolization
MeSH Terms: conditions — Vein of Galen Malformations; Vein of Galen aneurysm | interventions — Embolization, Therapeutic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vein of Galen malformation: All patients treated at Erasme hospital for a vein of Galen malformation.
  Interventions: Procedure: embolization therapy

INTERVENTIONS:
Procedure: embolization therapy — Embolization in the neuroradiological department is the Golden Standard for the treatment of vein of Galen malformations.

SUMMARY:
1. Foundations of the clinical research project:

   Vein of Galen vascular malformations are a group of rare cerebral vascular malformations with complex anatomy and severe clinical consequences. The pathology consists of direct communications between small intracerebral arteries and veins without the presence of capillaries. The result is a vascular malformation with low resistance and high flow, a lesion that will evolve during fetal development into aneurysmal dilatation.

   These lesions evolve towards rupture, but due to the high flow rate through these malformations, children very quickly develop cardiac decompensation (high-output failure). Treatment must be rapid, often on the first day of life. The technique currently used is iterative embolization. General anaesthesia is required for this procedure. However, neonatal anesthesia in children with cardiac decompensation and pulmonary hypertension poses major challenges for the anesthesia team. A high percentage of these patients require a short stabilization period with management of cardiac decompensation and pulmonary hypertension, most often by continuous milrinone infusion.

   Hôpital Erasme is a reference center for the management of vein of Galen malformations. In this work, we propose to analyze all cases of children with veins of Galen malformations managed by the interventional neuroradiology department.
2. Objectives of the clinical research project:

   2.1 Main objective:

   Description of cerebral lesions as described by angiography. Details of anesthetic management with all anesthetic drugs, details of cardiac management. Details of ventilatory management, intubation duration required.

   Description of embolization outcome. Description of the neurological and cardiac outcome.

   2.2 Secondary objectives:

   Possibly, depending on the number of patients, attempt to identify factors predictive of poor outcome.
3. Methodology of the clinical research project:

   We will carry out a retrospective analysis of the records of all patients who have been managed at Erasme for vein of Galen-type malformation. Activity began ± in 2011, and we will produce a listing of all patients from 2010 to August 2024. From this listing, obtained by the radiology department, we will collect data from the patients computer files.
4. Design of the clinical research project:

   This is a retrospective study based on file analysis.
5. Participants:

All patients treated at Erasme for a vein of Galen malformation. We will check the file to ensure that the parents have not expressed any opposition to the use of the patient medical data.

ELIGIBILITY:
Inclusion Criteria:

- All patients treated at Erasme for a vein of Galen malformation

Exclusion Criteria:

- Opposition of parents to the use of medical data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated at Erasme for a vein of Galen malformation up to august 2024
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Neurological outcome | 28 days
  Neurological outcome after each embolization therapy will be recorded (%): No neurological deficit, minor neurological deficit, major neurological deficit

SECONDARY OUTCOMES:
Cardiac failure | 28 days
  Presence of cardiac failure before, during and after each embolization therapy will be recorded. (%)
Inotropic support | 28 days
  Inotropic support for heart failure will be recorded (%), as well as the type of inotropic agents used for treatment and maximum dosage.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- H.U.B - Hôpital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashida Y, Miyahara H, Sawada H, Mitani Y, Maruyama K. Anesthetic management of a neonate with vein of Galen aneurysmal malformations and severe pulmonary hypertension. Paediatr Anaesth. 2005 Jun;15(6):525-8. doi: 10.1111/j.1460-9592.2005.01471.x. PMID 15910357
- [Background] Sinha PK, Neema PK, Rathod RC. Anesthesia and intracranial arteriovenous malformation. Neurol India. 2004 Jun;52(2):163-70. PMID 15269462
- [Background] Mortazavi MM, Griessenauer CJ, Foreman P, Bavarsad Shahripour R, Shoja MM, Rozzelle CJ, Tubbs RS, Fisher WS 3rd, Fukushima T. Vein of Galen aneurysmal malformations: critical analysis of the literature with proposal of a new classification system. J Neurosurg Pediatr. 2013 Sep;12(3):293-306. doi: 10.3171/2013.5.PEDS12587. Epub 2013 Jul 26. PMID 23889354